CLINICAL TRIAL: NCT03940664
Title: CD160 Expression in Retinal Vessels is Associated With Retinal Neovascular Diseases
Acronym: NEOVASC-CD160
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2018Ao001
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Surgical Retinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neovascular group: patients with diabetic retinopathy, retinal vein occlusion complicated with iris rubeosis or neovascular glaucoma, ocular ischaemic syndrome, neovascular glaucoma secondary to any ocular event or iris rubeosis secondary to retinal detachment
  Interventions: Other: immunohistochemistry on Formalin fixed and paraffin embedded blocks
- non-neovascular group: patients without neovascular diseases or complications but who underwent events leading to eye surgery such as trauma, endophthalmitis, cellulitis, anterior perforation, corneal abscess or retinal detachment.
  Interventions: Other: immunohistochemistry on Formalin fixed and paraffin embedded blocks

INTERVENTIONS:
Other: immunohistochemistry on Formalin fixed and paraffin embedded blocks

SUMMARY:
The aims of this study were

* to analyze CD160 expression in both normal and pathological eyes from human adults
* to evaluate association between CD160 presence on endothelial cells from blood vessels and retinal vascular disease

DETAILED DESCRIPTION:
Anti-angiogenic agents stand first in the treatment of neovascular diseases of the retina. Intravitreal injections of anti-Vascular Endothelial Growth Factor (VEGF) agents have emerged over the past decade as the first line of treatment in some neovascular diseases of the retina. Nevertheless, anti-VEGF therapies suffer some limitations, among which a short time to recurrence (1 week to 3 months) of retinal neovascularization and an eroding biological effect after prolonged use and.

CD160 appeared in several experimental studies as a marker of activated endothelial cells, suggesting it could represent a promising target for novel anti-angiogenic.

ELIGIBILITY:
inclusion criteria :

* Patients with retinal surgery
* Patients who agree to participate to the study
* Major patient

exclusion criteria :

* Patient under law protection
* Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with surgical retinal
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
CD160 staining intensity score | Day0
  Formalin fixed and paraffin embedded blocks were used for immunohistochemistry using CD160.
  The immunolabelling was evaluated independently by 2 observers (CBR, AH) blinded to clinical data. The staining intensity (0: absent, 1: faint, 2: moderate, 3: strong) was assessed for CD160 immunolabelling.

SECONDARY OUTCOMES:
CD105 staining intensity score | Day0
  Formalin fixed and paraffin embedded blocks were used for immunohistochemistry using CD105.
  The immunolabelling was evaluated independently by 2 observers (CBR, AH) blinded to clinical data. The staining intensity (0: absent, 1: faint, 2: moderate, 3: strong) was assessed for CD105 immunolabelling.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Henry A, Boulagnon-Rombi C, Menguy T, Giustiniani J, Garbar C, Mascaux C, Labrousse M, Milas C, Barbe C, Bensussan A, Durlach V, Arndt C. CD160 Expression in Retinal Vessels Is Associated With Retinal Neovascular Diseases. Invest Ophthalmol Vis Sci. 2018 Jun 1;59(7):2679-2686. doi: 10.1167/iovs.18-24021. PMID 29860454